CLINICAL TRIAL: NCT01973166
Title: Randomized, Split-tattoo Study Comparing Safety and Efficacy of Picosecond and Nanosecond Q-switched Nd:YAG Lasers for Tattoo Removal
Brief Title: Study of Picosecond and Nanosecond Q-switched Lasers for Tattoo Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-13-TPS04
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Tattoo Removal
Keywords: Tattoo Removal; Q-switched laser; Nd:YAG laser; Nanosecond laser; Picosecond laser; Laser therapy; Tattoo; pulsed-laser; laser treatment; remove tattoo; tattoo clearing; tattoo lightening; tattoo lighten

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Picosecond Q-switched Laser Treatment (Experimental): Picosecond Q-switched Nd:YAG (1064 nm and 532 nm) laser
  Interventions: Device: Picosecond Q-switched Laser Treatment
- Nanosecond Q-switched Laser Treatment (Active Comparator): Nanosecond Q-switched Nd:YAG (1064 nm and 532 nm) laser
  Interventions: Device: Nanosecond Q-switched Laser Treatment

INTERVENTIONS:
Device: Picosecond Q-switched Laser Treatment
  Arms: Picosecond Q-switched Laser Treatment
Device: Nanosecond Q-switched Laser Treatment
  Arms: Nanosecond Q-switched Laser Treatment

SUMMARY:
The purpose of this study is to compare the investigational medical grade laser device to a marketed medical grade laser device for effectiveness in lightening or clearing unwanted tattoos. This study will also compare any side effects from treatment with the devices.

DETAILED DESCRIPTION:
This is a two center study to evaluate the Cutera RF system. Subjects will be treated on the abdomen and / or flanks areas and / or saddle bag (upper lateral thigh, lateral hip and lower buttocks).

The objective of this study is to evaluate the thermal and histological changes observed in the subcutaneous tissue following RF exposure.

ELIGIBILITY:
Inclusion Criteria:

* Females or Males, 18 to 65 years of age (inclusive)
* Fitzpatrick Skin Type I - IV (Appendix 3)
* Tattoos containing black/blue ink alone or in combination with other colors
* Target tattoos older than 1 year
* Presence of tattoos equal or greater than 2 square inches, not to exceed 12 square inches
* Must be able to read, understand and sign the Informed Consent Form
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions
* Wiling to cover tattoos with a bandage or clothing; and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area starting 2 to 4 weeks before the treatment and/or every day for the duration of the study, including the follow-up period
* Willing to use hydroquinone approximately 4 weeks pre-treatment and post- treatment if required
* Willingness to have digital photographs taken of the treated area
* Agree not to undergo any other procedure(s) for the tattoo removal during the study
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study

Exclusion Criteria:

* Participation in a study of another device or drug within 6 months prior to enrollment or during the study
* Prior treatment for tattoo removal in the target area, e.g., with q-switched laser, IPL, dermabrasion, electrocautery, cryotherapy
* History of allergic reaction to pigments following tattooing
* Presence of double tattoo in the treatment area
* History of allergy to local anesthetics
* History of allergy to topical antibiotics
* History of malignant tumors in the target area
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles
* Pregnant and/or breastfeeding
* Having an infection, dermatitis or a rash in the treatment area
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension
* Suffering from coagulation disorders or taking prescription anticoagulation medications
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications
* History of vitiligo, eczema, or psoriasis
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma
* History of seizure disorders due to light
* Any use of medication that is known to increase sensitivity to light, such as tetracycline
* History of herpes simplex and/or herpes zoster (shingles)
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation
* Systemic use of corticosteroid within 12 months of study participation
* Use of oral isotretinoin within 12 months of study participation and topical use of isotretinoin within 6 months on the treated area
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study
* Current smoker or history of smoking within 6 months of study participation
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Apfelberg, Principal Investigator — Study Principal Investigator
Locations (1):
- Brisbane, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: halves of tattoo
Groups:
- All Study Participants: Subject tattoos were divided into 2 portions for assignment into 2 treatment arms: active control arm and treatment arm. One tattoo portion was treated with the Cutera Investigational picosecond Q-Switched Nd:YAG laser and the other tattoo portion with a comparator nanosecond Q-switched Nd:YAG laser
Period: Overall Study
Arm/Group | All Study Participants
Started | 42; 84 halves of tattoo
Treatment With Cutera Investigational Picosecond Q-Switched Nd:YAG Laser | 42; 42 halves of tattoo
Treatment With Comparator Nanosecond Q-switched Nd:YAG Laser | 42; 42 halves of tattoo
Completed | 41; 82 halves of tattoo
Not Completed | 1; 2 halves of tattoo

BASELINE CHARACTERISTICS:
Groups:
- Picosecond and Nanosecond Q-Switched Laser Treatment: Picosecond and Nanosecond Q-Switched Laser Treatment (532 nm and 1064 nm)
Arm/Group | Picosecond and Nanosecond Q-Switched Laser Treatment
Number analyzed (Participants) | 42
Age, Continuous [Mean (Full Range); unit: years] | 34 [20 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 2
  Unknown or Not Reported | 15

OUTCOME MEASURES:

1. Primary Outcome: Tattoo Clearing at 6 Weeks Post-final Laser Treatment for Each Treatment Arm as Assessed by Blinded Reviewers.
Description: Physician's Global Assessment Scale: 0 (min) - 4 (max) Higher scores represent better tattoo clearing 4 = Very Significant Clearing (> 75%) 3 = Significant Clearing (51 - 75%) 2 = Moderate Clearing (26 - 50%)
  1 = Mild Clearing (5 - 25%) 0 = No Change (< 5%)
Time Frame: 6-weeks post-final treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Picosecond Q-switched Laser Treatment: Picosecond Q-switched Nd:YAG (1064 nm and 532 nm) laser
  Picosecond Q-switched Laser Treatment
- Nanosecond Q-switched Laser Treatment: Nanosecond Q-switched Nd:YAG (1064 nm and 532 nm) laser
  Nanosecond Q-switched Laser Treatment
Arm/Group | Picosecond Q-switched Laser Treatment | Nanosecond Q-switched Laser Treatment
Number analyzed (Participants) | 41 | 41
score on a scale | 2.54 [2.13 to 2.94] | 2.17 [1.77 to 2.57]

2. Secondary Outcome: Comparison of Subject Discomfort (Pain) Between Treatment and Active Control Treatment Arms During Treatment
Description: Numeric Pain Rating Scale (Min=0; Max=10) Higher scores mean worse outcome
Time Frame: During treatment, approximately 10 minutes
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Picosecond Q-switched Laser Treatment | Nanosecond Q-switched Laser Treatment
Number analyzed (Participants) | 42 | 42
score on a scale | 4.1 [0.5 to 9] | 4.4 [0 to 9]

ADVERSE EVENTS:
Groups:
- Picosecond Q-Switched Laser Treatment: Picosecond Q-Switched Laser Treatment (532 nm and 1064 nm)
- Nanosecond Q-Switched Laser Treatment: Nanosecond Q-Switched Laser Treatment (532 nm and 1064 nm)
Arm/Group | Picosecond Q-Switched Laser Treatment | Nanosecond Q-Switched Laser Treatment
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 42/42 | 42/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Picosecond Q-Switched Laser Treatment (N=42) | Nanosecond Q-Switched Laser Treatment (N=42)
Pinpoint Bleeding (Skin and subcutaneous tissue disorders) | 32 | 20
Edema (Skin and subcutaneous tissue disorders) | 42 | 42
Erythema (Skin and subcutaneous tissue disorders) | 42 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No